CLINICAL TRIAL: NCT01929564
Title: Broccoli and Vascular Health Study
Acronym: BASH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Quadram Institute Bioscience (Other)
Collaborators: Biotechnology and Biological Sciences Research Council (Other); Technology Strategy Board, United Kingdom (Other); Monsanto Company, LLC (Industry); University of Reading (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: IFR01/2012
Record Dates: First submitted 2013-03-27; First posted 2013-08-28 (Estimated); Last update posted 2014-07-29 (Estimated); Status verified 2014-07

CONDITIONS: Cardiovascular Diseases
Keywords: cardiovascular disease; risk factor; broccoli; GST; blood pressure; Total cholesterol
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Beneforte broccoli (Active Comparator): Four x 100g portions of Beneforte broccoli will be consumed each week for twelve weeks, on top of the participants habitual diet.
  Interventions: Other: Beneforte broccoli
- Parthenon broccoli (Placebo Comparator): Four x 100g portions of Parthenon broccoli will be consumed each week for twelve weeks, on top of the participants habitual diet.
  Interventions: Other: Parthenon Broccoli

INTERVENTIONS:
Other: Beneforte broccoli — Four x 100g portions of Beneforte broccoli will be consumed each week for twelve weeks, on top of the participants habitual diet
  Arms: Beneforte broccoli
Other: Parthenon Broccoli — Four x 100g portions of Parthenon broccoli will be consumed each week for twelve weeks, on top of the participants habitual diet
  Arms: Parthenon broccoli

SUMMARY:
The participants of this study will be men & women ≥50 years who are deemed to have a 10-30% risk of developing CVD over the next 10 years. Their risk will be calculated using the Joint British Societies 2 (JBS2) guidelines on the prevention of CVD in clinical practise algorithm. This takes into account the participants age, sex, cholesterol values, blood pressure,family history and their ethnicity (SE Asian or not). The participants will be randomly assigned to one of two groups with the aid of a computer program called "minim" which uses their age, sex, BMI and smoking status to determine which broccoli each participant will consume on the intervention.

Each participant will consume 4 x 100g of their assigned broccoli, each week for 12 weeks on top of their normal diet. They will be allowed to eat the broccoli whenever they want during the week, but will be asked to note down when they eat it. A steamer will be provided so participants can cook their broccoli for the required 4-5 minutes. Participants will be asked to keep two diet diaries during their time on the intervention, one before they start the intervention and one towards the end. Blood samples and urine will also be collected, pre and post intervention, for the analysis of biomarkers of CVD.

This is joint project based at two sites, the Institute of Food (IFR) Research in Norwich and the University of Reading(UoR), in Reading. Samples from the participants at both sites will be analysed at IFR, UoR and companies in the United States.

DETAILED DESCRIPTION:
This intervention will take place at two independent sites, The Institute of Food Research's Human Nutrition Unit (HNU)in Norwich and the Hugh Sinclair Human Nutrition Unit (HSU), at the University of Reading. The participants recruited from Norwich and Reading will solely attend the unit in their area and the paper work has been written to reflect this i.e.separate participant information sheets (PIS). In addition to the tests carried out at both sites, the Reading cohort will also undergo additional vascular tests, also reflected in the PIS. Despite the sites being independent, 96 participants will be recruited across both sites, with the possibility of uneven numbers from each site making up the final number.

The purpose of this study is to assess whether diet can affect an individuals chances of developing CVD, as it is one of the biggest killers in the UK. We are particularly interested in participants who have a 10%-30% risk of developing CVD. We are able to assess a person's risk with the help of the Joint British Societies 2 guidelines on the prevention of cardiovascular disease, cardiovascular disease risk prediction chart. These charts take a number of parameters we obtain from the participant, their age, sex, total cholesterol concentration, systolic blood pressure (BP), body mass index (BMI), serum high density lipoprotein concentration, their smoking status and diabetes status and put them into an algorithm. The result is a risk score out of 100, of a person developing CVD over the next 10 years.

The study will be conducted over two sites, Reading and Norwich, with a principal investigator assigned to each site. The total number of participants recruited over both sites will be 96. It may be that uneven numbers are recruited over the two sites e.g. 46 at one and 50 at another however regardless of the number at each site, 48 participants will be assigned to each of the two groups. One group will consume 400g of the commercially available high glucosinolate Beneforté® broccoli each week for 12 weeks and the other will consume 400g of a standard broccoli, Parthenon for 12 weeks.

As we are assessing the effect of diet on CVD risk, our participants will be screened initially. Their urine will be tested (urine dipstick test), their height, weight, waist and hip measurements, BMI, BP will be measured and questions linked to lifestyle choices (alcohol consumption, smoking status and physical activity) will be asked. A separate section pertaining to women's health will also be present on the questionnaire.

All participants will be asked to give written informed consent before they can participate in the intervention study. The Reading cohort will be sent a copy of the consent and medical declaration forms to read through at home. The forms sent to the homes will be clearly distinguishable from the real forms as they will have the watermark with "SAMPLE" written across them.

CVD risk assessment calculator This calculator will be used once the results of the screening are known. A program devised by the University of Manchester will be used to calculate the risk our participants have of developing CVD over the next 10 years. This program is based on the Joint British Societies 2 guidelines on the prevention of CVD risk prediction charts. For the purposes of this study we would like our participants to fall into the 10%-30% risk category as most literature suggests people in this range may benefit from dietary change, without the need for medication, in the most part. The CVD risk scores will be sent to the participants GP and we will continue to advise our participants to discuss the results with their GPs if they score >10%.

Genotyping There is evidence to suggest that a person's genetic make-up may affect the way isothiocyanates (ITCs), one of the active components of broccoli, work. Of the 30,000 genes found in humans a group of genes associated with the protein glutathione S-transferase M1 (GSTM1) has been shown to affect ITCs after consumption and has been implicated in CVD. There is evidence to suggest that individuals with a deletion in GSTM1 breakdown the glucosinolate, from which the ITC sulforaphane is derived, differently to individuals that have the gene. We also know that glutathione S-transferase theta-1 (GSTT1) may also be involved in reducing the likelihood of developing CVD.

Along with the GST gene family and their association with cruciferous vegetables, there are a number of other genes that have been implicated in CVD itself. These include genes associated with lipid metabolism, thrombosis, leukocyte adhesion and nitric oxide production and thus blood vessel dilation. This is by no means an exhaustive list and will therefore remain open to other viable candidates.

Vascular measurements As we age, our arteries stiffen which causes an increase in the demands of the heart and an increase in blood pressure. This increase in BP can dramatically increase the risk of heart attack, stroke and heart failure. Arterial stiffness has also been associated with many of the common risk factors associated with CVD such as age, high blood pressure, smoking, cholesterol levels and obesity, but importantly, arterial stiffness has been shown to be an independent predictor of CVD in a large section of society.

There are many ways in which arterial stiffness can be assessed. We will be looking at blood pressure, which will be very familiar to most participants in our age range (over 50yrs of age). The only difference being that the participant will wear a cuff for an hour and readings will be collected every ten minutes.

Another method will be Pulse Wave Analysis (PWA), where a probe will be held against the neck and the upper thigh to take the measurements for up to a minute at a time. As participants may not be wholly familiar with this technique, it is hoped that a short video clip could be shown on a laptop or diagrams/photographs of the technique will be discussed with the participant at screening.

Restricted conditions prior to study day Before the study day the participants will be asked to abstain from a number of activities. This will be clearly stated in the PIS.

These include:

1. No alcohol or caffeine for 24 hours before the study day. Participants who consume a lot of caffeine will be advised that they may suffer from headaches. They will be asked to tell the study scientist if they needed to take any medication as a consequence.
2. Low fat meal to be consumed the night before the study day. Participants will be asked to eat a low fat meal from a selected list that we give them. We will ask that the meal is consumed before 10pm, as the participants will then have to fast for their study day.
3. Fasting for at least 8 hours. Participants will need to fast for at least 8 hours. This means that they won't be able to eat or drink anything, apart from water during this time. They can drink as much water as they feel they need.
4. No heavy exercise the morning of their study day. Participants will be asked not to engage in any vigorous exercise the morning of their study day. This will be defined as any activity that causes an increase in heart rate, panting and/or sweating. A participant who normally cycles will be asked not to on the morning of their study day.
5. No smoking an hour before their study day measurements. All participants that smoke will be asked to abstain from smoking at least an hour before their study day. We would also ask that they avoid all passive smoking.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged ≥ 50 years will be recruited onto the study using the JBS 2 cardiac risk assessor calculator.

Scores of 10%-30% will be acceptable for participation in the study.

Exclusion Criteria:

* Those unable to give written informed consent
* Those unwilling to provide GP details
* Those already consuming Beneforté ® broccoli, unless they are willing to discontinue consumption for 8 weeks prior to starting the study.
* Diagnosed diabetics
* Fasting glucose >7mmol/L (WHO guidelines for diabetics)
* Blood pressure <90/50 or 95/55 if symptomatic; >160/100
* Chronic kidney disease
* BMI <20
* BMI >40
* Fasting total cholesterol > 8.0mmol/L
* Fasting glucose >7mmol/L (WHO guidelines for diabetics)
* Blood pressure <90/50 or 95/55 if symptomatic; >160/100
* Chronic kidney disease
* BMI <20
* BMI >40
* Fasting total cholesterol > 8.0mmol/L
* Haemoglobin Men <13.8g/dL (8.56mmol/L) Women <12.1g/DL (<5.51mmol/L)
* Peri-menopausal women (defined as : when there is a change in menses)
* Women on HRT for less than one year
* Women who are pregnant or breastfeeding
* Those taking self-prescribed aspirin for cardiovascular reasons
* All those taking blood pressure medication
* Those on any lipid lowering therapies such as statins, bile acid sequestrants, cholesterol absorption inhibitors and nicotinic acid
* Those on regular medication for hypercoagulation and inflammatory conditions e.g. corticosteroids and asthma (intermittent use of an inhaler will be discussed on an individual basis)
* Those on glucose lowering medications
* Those who have ever suffered a cardiovascular event such as stroke, myocardial infarction or trans ischemic attacks
* Peripheral vascular disease including Claudication
* Consumption of fish oil supplements (unless participant is willing to discontinue their use 8 weeks prior to the start of the intervention- all other supplements with be dealt with on an individual basis)
* Parallel participation in another research project which involves dietary intervention and/or sampling of blood
* Any person related to or living with any member of the study team
* Participation in another research project which involves blood sampling within the last four months unless the total blood from both studies (including this one) does not exceed 470mL)
* Those who have donated or intend to donate blood within 16 weeks of the first and last study samples
* Gastrointestinal disease (excluding hiatus hernia) unless symptomatic or study intervention/procedure is contraindicated
* Going on holiday for more than two weeks during the intervention
* Those undergoing any on-going GP investigation

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2012-07; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure is to assess the change in CVD risk after a 12 week broccoli intervention by assessing the change in concentration of LDL-cholesterol on which the power calculation was based. | Baseline and 12 weeks
  The LDL cholesterol concentration (mmol/L) will be measured before and after a 12 week intervention with broccoli, using a Instrumentation Laboratories kit for use on an ILAB auto analyser.

SECONDARY OUTCOMES:
To assess the effects of the broccoli intervention clinical biomarkers of CVD. The effect of the intervention on arterial stiffness will also be measured on a sub section of the total cohort (measurements carried out on the Reading cohort). | Baseline and 12 weeks.
  The clinical biomarkers include, hs-CRP (mg/L), NEFAs(mg/dL), Plasma NO(umol/L), hs-IL6(pg/mL), TNF-α(pg/mL), ox LDL(umol/L), IL-1beta(pg/L), PCOOH(pmols/L), F-2 isoprostanes (mg/mL/mg creatine) and 8-OHdG (ng/mL).
  The effect of the intervention on arterial stiffness on a sub section of the cohort (Reading cohort)will also be measured. The first measurement will be Pulse wave velocity (m/sec); the 2nd measurement will be Laser Doppler Imaging with iontophoresis (perfusion units(area under the blood flow.time curve)).

OTHER OUTCOMES:
To determine the genotype of the participants. | Measurements will be made using either a pre or post intervention sample
  DNA samples from all participants will be genotyped for PAPOLG (NM_022894.3) rs11687951, rs28459296 and rs7579240 and GSTM1 genotype using predesigned Invitrogen TaqMan® Assays according to manufacturers' instructions.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Mithen, Professor, Study Director — Quadram Institute Bioscience
Locations (2):
- United Kingdom (2):
  - University of Reading, Reading, Berkshire
  - Institute of Food Research, Norwich, Norfolk